CLINICAL TRIAL: NCT00255333
Title: A Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Weekly Intravenous INNO-105 in Adult Patients With Advanced Solid Malignancies
Brief Title: INNO-105 in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development of this compound was discontinued.
Sponsor: Innovive Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-105-901
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — Enkephalin, Methionine

INTERVENTIONS:
Drug: INNO-105

SUMMARY:
The safety, tolerability and pharmacokinetics of INNO-105, an investigational anticancer drug, are being studied in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of a solid malignancy (patients may have either measurable or nonmeasurable disease).
2. Be ≥18 years old.
3. Not eligible for effective therapy likely to provide clinical benefit.
4. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
5. Acceptable pretreatment clinical laboratory results.
6. Life expectancy of greater than 12 weeks.

Exclusion Criteria:

1. Have received previous treatment with INNO-105.
2. Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
3. Are pregnant or lactating.
4. Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
5. Have received any chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational, within 2 weeks of treatment in this study.
6. Have not recovered from acute toxicity of all previous therapy prior to enrollment.
7. Have symptomatic or untreated central nervous system (CNS) metastases.
8. Have a susceptibility to hypotension, bradycardia, and/or hypopnea, such as patients with known coronary heart disease, arrhythmias, cerebral vascular disease, and chronic obstructive airways disease (CO2-retaining).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-11; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Cunningham, MD, Principal Investigator — Mary Crowley Medical Research Center; Edward Sausville, M.D., Ph.D., Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Mary Crowley Medical Research Center, Dallas, Texas